CLINICAL TRIAL: NCT05171569
Title: Post Discharge After Surgery Virtual Care With Remote Automated Monitoring Technology-3 (PVC-RAM-3) Trial
Brief Title: Post Discharge After Surgery Virtual Care With Remote Automated Monitoring Technology-3 Trial
Acronym: PVC-RAM-3
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: v2.0_2025-01-25
Record Dates: First submitted 2021-12-10; First posted 2021-12-29 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Surgery
Keywords: Virtual care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Care with Remote Automated Monitoring (Experimental): Patients randomized to the PVC-RAM-3 intervention will take biophysical measurements with the RAM technology, complete a daily recovery survey, complete video visits with a virtual care clinical team, and take wound photos during the 14 days after discharge. If the patient's RAM measurements exceed predetermined thresholds, the patient reports specific symptoms (e.g., shortness of breath), a drug error is identified, or the virtual nurse has concerns about the patient's health that they cannot resolve, the virtual nurse will escalate care to a pre-assigned and available physician.
  Interventions: Device: Virtual care with remote automated monitoring (RAM)
- Standard Care (No Intervention): Standard post surgical care per treating institution.

INTERVENTIONS:
Device: Virtual care with remote automated monitoring (RAM) — Use of Cloud Diagnostics connected health kit for at home monitoring with virtual clinical from nursing and perioperative physician team.
  Arms: Virtual Care with Remote Automated Monitoring

SUMMARY:
The Post discharge after surgery Virtual Care with Remote Automated Monitoring technology (PVC-RAM)-3 Trial is a multicentre, parallel group, superiority, randomized controlled trial to determine the effect of virtual care with remote automated monitoring (RAM) technology compared to standard care on length of index hospital stay and use of acute hospital care (composite of hospital readmission and emergency department visit) after randomization, in adults who have undergone elective non cardiac surgery. Secondary outcomes at 30 days after randomization include: 1) hospital re-admission; 2) emergency department visit; 3) medication error detection;4) medication error correction; 5) surgical site infection; and 6) days in hospital. Additional secondary outcomes are pain of any severity, and moderate-to-severe pain assessed at 15 and 30 days after randomization. The investigators will also assess optimal management of long-term health by evaluating among patients with atherosclerotic disease and current smokers whether patients are taking classes of efficacious medications at 30 days.

ELIGIBILITY:
Inclusion Criteria:

1. are ≥18 years of age;
2. are undergoing inpatient elective noncardiac surgery with an expected length of hospital stay ≤3 days after surgery; and
3. provide informed consent to participate.

Exclusion Criteria:

1. are unable to communicate with research staff, complete study surveys, or undertake an interview using a tablet computer due to a language barrier or a cognitive, visual, or hearing impairment; or
2. reside in an area without cellular network coverage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Index hospital length of stay | 30 Days post randomization
  Length of stay from randomization until discharge from the index hospitalization (measured in days and hours)
Acute hospital care (composite of hospital readmission and emergency department visit) | 30 Days post randomization
  Acute-hospital care is a composite outcome of hospital re-admission and emergency department visit, which includes urgent-care centre visit.

SECONDARY OUTCOMES:
Hospital readmission | 30 days post randomization
  Patient admission to an acute-care hospital.
Emergency department visit (includes urgent care centre visit) | 30 days post randomization
  Patient visit to an emergency department, which includes urgent-care centre visit.
Medication error detection | 30 days post randomization
  Medication errors include mistakes in medication prescribing, transcribing, dispensing, administering, or monitoring due to preventable events or actions taken by a patient, caregiver, or healthcare worker. Medication errors include: drug omission (i.e., patient did not take a drug they were supposed to take), drug commission (i.e., patient taking a drug they were not supposed to take), duration error, dosing error, frequency error, route error, and timing error. We will record all drug errors identified.
Medication error correction | 30 days post randomization
  Any medication error that is corrected.
Surgical site infection | 30 days post randomization
  Surgical site infection is an infection that occurs within 30 days after randomization and involves the skin, subcutaneous tissue of the incision (superficial incisional), or the deep soft tissue (e.g., fascia, muscle) of the incision (deep incisional).
Days in hospital | 30 days post randomization
  Days in hospital
Level of pain and pain related interference in recovery | 15 and 30 days post randomization
  Pain intensity and related interference with usual daily activities, will be measured via the Brief Pain Inventory-Short Form (BPI-SF).4 The BPI-SF includes four 11-point numeric rating scales (NRS) of pain intensity, which measure "average", "least", and "worst" pain intensity in the past 24 hours (hrs.), respectively, as well as pain intensity "now" (0= no pain, 10= pain as bad as you can imagine). The BPI-SF interference subscale will also be used, which measures the degree to which pain interferes with general activity, mood, walking, work, relations with others, sleep, and enjoyment of life (NRS for each item; 0=does not interfere, 10=completely interferes). A total interference score is determined by calculating the sum of these 7 items. The BPI-SF has strong psychometric properties with well-established reliability and validity across divergent surgical groups. Moderate to severe pain is defined by a score of ≥4/10 on a standard numeric rating scale (NRS) for pain.
Optimization of medications for long-term health | 30 days post randomization
  Among patients with atherosclerotic disease, we will also assess optimal pharmacological management based upon whether patients are taking 0, 1, 2, or 3 of the following classes of efficacious medications at 30 days (i.e., an antiplatelet or anticoagulant drug; an angiotensin-converting enzyme inhibitor or angiotensin-receptor blocker; and a statin). Among active smokers before surgery we will assess if patients are receiving pharmacological smoking cessation interventions at 30 days after randomization.

OTHER OUTCOMES:
Infection | 30 days post randomization
  Infection is defined as a pathologic process caused by the invasion of normally sterile tissue, fluid, or body cavity by pathogenic or potentially pathogenic organisms.
Re-operation | 30 days post randomization
  Re-operation refers to any surgical procedure undertaken for any reason (e.g., wound dehiscence, infection).
Composite of myocardial infarction, acute heart failure, and arrhythmia that results in acute hospital care | 30 days post randomization
  The diagnosis of myocardial infarction requires criteria meeting 4th universal definition of myocardial infarction.
  The definition of acute heart failure requires at least one of the following clinical signs (i.e., elevated jugular venous pressure, respiratory rales or crackles, crepitations, or presence of S3) with at least one of the following:
  1. radiographic findings of vascular redistribution, interstitial pulmonary edema, or frank alveolar pulmonary edema, OR
  2. heart failure treatment with a diuretic and documented clinical improvement.
  Any arrhythmia that results in patient presenting to an emergency department, which includes an urgent care centre visit or being admitted to hospital.
Death | 30 days post randomization
  All cause mortality
Health related quality of life (HRQoL) | 30 days post randomization
  HRQoL will be measured with the EQ-5D-5L instrument (https://euroqol.org/eq-5d-instruments/sample-demo) due to its increased sensitivity and validation in several countries including Canada.4 The EQ-5D-5L is also recommended in Canada5 to calculate the Quality Adjusted Life Years (QALYs) when conducting cost-effectiveness analyses.
Health services utilization-related costs | 30 days post randomization
  Data on hospital re-admission, length of stay, and healthcare utilization will be obtained from the Ontario Hospital Association Integrated Decision Support (IDS) database. IDS is a comprehensive platform with an integrated view of patient activity, allowing for access to health systems data for any patients enrolled. Data on costs of health service utilization will be obtained from the Ontario Case Costing Database.

CONTACTS AND LOCATIONS:
Overall Officials: Michael McGillion, PhD, Principal Investigator — McMaster University, Population Health Research Institute; PJ Devereaux, M.D, PhD, Principal Investigator — McMaster University, Population Health Research Institute
Locations (2):
- Canada (2):
  - Hamilton General Hospital, Hamilton, Ontario
  - Juravinski Hospital, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ofori S, McGillion MH, Borges FK, Ouellette C, Patel A, Conen D, Marcucci M, Wang MK, Park LJ, Bell C, Lounsbury J, Nagatani K, Tandon V, Wilkieson TJ, Wyne A, Harvey V, Harrison S, Nenshi R, Bogach J, Harlock J, Cadeddu M, Forbes S, Haider S, Mirza RD, Narang S, Reade CJ, Tushinski DM, Raut A, Raza S, Scott T, Adili A, Petch J, Devereaux PJ. Impact of Virtual Care With Remote Automated Monitoring on the Rate of Acute Hospital Care Post Discharge and Index Length of Hospital Stay: Protocol for the Post Discharge After Surgery Virtual Care With Remote Automated Monitoring Technology 3 (PVC-RAM-3) Trial. JMIR Res Protoc. 2025 Jun 2;14:e72672. doi: 10.2196/72672. PMID 40456137